CLINICAL TRIAL: NCT00742014
Title: The Assessment of Right Ventricular Contractility in Response to Sildenafil in Pediatric Patients With Pulmonary Arterial Hypertension
Brief Title: The Assessment of Right Ventricular Contractility in Response to Sildenafil
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: absorption of oral sildenafil not consistent
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000012265
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2016-04

CONDITIONS: Hypertension
Keywords: Pulmonary arterial hypertension; Pediatrics; Sildenafil; Catheterization; Right ventricular contractility
MeSH Terms: conditions — Hypertension; Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — One oral dose of Sildenafil (0.5 mg/kg) will be administered nia a nasogastric tube
  Other Names: Viagra

SUMMARY:
The primary objective of this study is to examine the effects of Sildenafil, administered during cardiac catheterization, on right ventricular contractility in children with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
The effectiveness of Sildenafil as a pulmonary vasodilator in children with heart disease was first reported in detail during cardiac catheterization and postoperatively in 2003. It is now used frequently for long-term treatment of children with pulmonary arterial hypertension at The Hospital for Sick Children and it is now a routine part of the hospital's testing protocol for all patients being evaluated for pulmonary hypertension in the cardiac catheterization laboratory.

The beneficial effects of Sildenafil in pulmonary hypertension are thought to result predominantly from relative vasodilatory and antiproliferative effects on the pulmonary vasculature. On the basis of early data showing lack of significant PDE5 expression in the normal heart, PDE5 was thought to be expressed in the coronary vessels but not in the human myocardium. Very recently, it was reported for the first time that PDE5 is markedly upregulated in hypertrophied right ventricular myocardium in humans and that in the rat PDE5 inhibition with Sildenafil increases contractility in hypertrophied right ventricular myocardium but not in normal right ventricle, which lacks PDE5 expression. The assessment of right ventricular contractility in humans is a challenge, but we have developed several techniques that are recognized as 'state of the art' assessment of right ventricular function.

The purpose of this study is to examine the effects of Sildenafil, which is routinely administered during cardiac catheterization to assess pulmonary vascular resistance, on right ventricular contractility in children with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Significant pulmonary arterial hypertension (mean pulmonary artery pressure > 25 mm Hg)
* Patients aged 4-18 years
* Routine cardiac catheterization clinically indicated for deciding therapeutic treatment
* Informed assent/consent from patient/parent

Exclusion Criteria:

* Suprasystemic pulmonary artery pressures
* Evidence of right heart failure
* History of ventricular arrhythmia
* Known vascular access arrhythmia
* Contraindication to Sildenafil
* Concurrent inotropic / PDE administration
* Other medical, psychological or social circumstances which complicate a regular participation in the study, and/or increase the risk for the patients themselves
* No consent/assent
* Pregnancy or unwillingness to comply with contraceptive advice

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Increase (% change) in endsystolic elastance of the right ventricle from baseline (in comparison to change in endsystolic elastance after inhaled NO) | 30 mins after Sildenafil adminsitration

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Redington, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada